CLINICAL TRIAL: NCT04453670
Title: A Prospective Observational Autopsy Study of Neuropathology in Adults Intensive Care Unit Patients With COVID 19
Brief Title: Neuropathology in Adults Intensive Care Unit Patients With COVID 19
Status: Completed | Type: Observational
Sponsor: University of Versailles (Other)
Responsible Party: Principal Investigator, Djillali Annane, Professor in intensive care medicine, University of Versailles
Other Study IDs: Obs2020
Record Dates: First submitted 2020-05-15; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: COVID 19
Keywords: autopsy; coronavirus; brain; inflammation
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Inflammation | interventions — Autopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma cerebrospinal fluid brain parenchyma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 non-survivors: ICU adults who died from severe COVID-19 and in whom autopsy could be performed
  Interventions: Procedure: autopsy

INTERVENTIONS:
Procedure: autopsy — autopsy

SUMMARY:
This is a single center observational autopsy study, conducted during the first wave of the coronavirus disease (COVID-19) pandemic in France. The main objective is to evaluate brain damages in patients who died from COVID-19 to inform the cause of death. Investigations include macroscopic and histology examinations, and virology analyses.

DETAILED DESCRIPTION:
Setting: academic center designed as a referral center for patients with COVID-19 Design: single center observational autopsy study Participants: intensive care unit (ICU) adults who died from confirmed COVID-19 during the first wave of the pandemic in France.

Oversight: As per legal health authority requirement only patients with suspected or confirmed severe acute respiratory syndrome (SARS)- related to coronavirus 2 infection were admitted to the ICU. The department of pathology and forensic medicine is allowed by legal authority to perform autopsy of non-survivors from COVID-19 to inform the cause of death as per ministerial decree of July 12 2017 and March 28, 2020. In this context, of autopsy for medical purpose and public interest there is no requirement for institutional review board submission. However, consent from patients legal representative or closest relatives is required for autopsy.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* admitted to the ICU
* confirmed COVID-19
* died during ICU stay

Exclusion Criteria:

* refusal from patient's legal representative or closest relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to the ICU for severe COVID-19 and who died during their ICU stay and for whom family consent was obtained for performing autopsy
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
detection of severe acute respiratory syndrome related to coronavirus-2 in brain tissues | From death up to five days
  Specimens treatments Genome detection by real-time reverse transcriptase-polymerase chain reaction and viral culture Next generation sequencing Specimen RNA pre-treatment and evaluation MinION sequencing
quantification of inflammation, necrosis and hemorrhage in different brain areas | From death up to five days
  The left hemisphere will be fixed in 10% buffered formalin. Multiple fresh samples will be acquired from different areas of the right hemisphere for freezing. For each frozen sample, a mirror sample of formalin-fixed paraffin-embedded tissue will be taken from the left hemisphere. Samples were fixed with 3.6% glutaraldehyde and embedded in plastic for electron microscopy. Paraffin sections cut to 3-µm thickness will be stained with hematoxylin and eosin stain. Immunohistochemistry will be performed with Clusters of Differentiation 3,4, 20, 68, 138, and glial fibrillary acid protein antibodies on automated immunostainer. Slides will be scanned and analyzed. Electron microscopy will be performed and images will be acquired.

CONTACTS AND LOCATIONS:
Overall Officials: djillali annane, Study Chair — University Versailles SQY Unversité Paris Saclay
Locations (1):
- Hôpital Raymond Poincaré, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided
all individual patient data will be available upon request to the study official and after signing a data sharing agreement immediately after publication in a peer-reviewed journal